CLINICAL TRIAL: NCT03815136
Title: The Effectiveness of Improved Use of Chewing Gum in Influencing Capsule Endoscopy Transit Time: A Prospective Randomized, Controlled Pilot Study
Brief Title: The Effectiveness of Chewing Gum in Influencing Capsule Endoscopy Transit Time
Acronym: CGCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CG-HuY-1901
Record Dates: First submitted 2019-01-20; First posted 2019-01-24 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Gastric Transit Time; Small-bowel Transit Time
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: Patients aged 16-80 years who were scheduled to undergo the small bowel capsule endoscopy(SBCE).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patients were instructed not to tell the endoscopist or the investigators about whether or not they used chewing gum before, during, or after the SBCE procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chewing Gum (Active Comparator): The subject group will chew sugarless chewing gum for a specific amount of time while undergoing capsule endoscopy. Subjects chewed one piece of gum for approximately 15 min every 30 min at the first hour of the examination.
  Interventions: Other: Chewing Gum
- Control (Placebo Comparator): The control group will not chew chewing gum while undergoing capsule endoscopy.
  Interventions: Other: Control

INTERVENTIONS:
Other: Chewing Gum — Patients of CG group chewed one piece of sugarless gum for approximately 15 min every 30 min at the first hour of the examination.
  Arms: Chewing Gum
Other: Control — The control group will not chew chewing gum while undergoing capsule endoscopy
  Arms: Control

SUMMARY:
The purpose of this study is to determine the effect of chewing gum, during the first one hour of examination in patients undergoing CE for GTT and SBTT time and the proportion of cases with complete small bowel examination and gastroscopy intervention.

DETAILED DESCRIPTION:
The participants will include patients who need to a capsule endoscopy (CE) in this unit. The investigators will include 200 participants who had a CE at our centre based on the gastric transit times. These will be randomly divided into two groups. The participants (chew chewing gum) and the controls (do not chew chewing gum).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years and <80 years old presenting for capsule endoscopy. Obtained of written informed consent before the procedure.

Exclusion Criteria:

* Patients on motility enhancing and/or slowing drugs(narcotics/prokinetics) should stop these at least 7 days prior to the procedure.
* Patients, who have proven or suspected obstruction of the bowel.
* Patients, who have had prior small bowel and/or gastric surgery.
* Patients, who have a dysphagia prohibiting.
* Patients with diabetes mellitus and/or hypo-/hyper-thyroidism.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
gastric transit time | 1 hour
  the time interval between the first gastric image and the first duodenal image
small bowel transit time | 8 hour
  The time interval between the first duodenal images and the first caecal image

SECONDARY OUTCOMES:
Completion rate | 9 hours
  the capsule reaching the caecum
Diagnostic yield | 9 hours
  the total number of positive (diagnostic and suspicious) findings
Intervention rate | 1 hours
  Gastroscopy intervention after capsule endoscopy not through pylorus within 1hour

CONTACTS AND LOCATIONS:
Overall Officials: Bin Lv, M.D., Principal Investigator — First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data sharing will be consider after study

REFERENCES:
- [Derived] Huang L, Hu Y, Chen F, Liu S, Lu B. Effectiveness of Improved Use of Chewing Gum During Capsule Endoscopy in Decreasing Gastric Transit Time: A Prospective Randomized Controlled Study. Front Med (Lausanne). 2021 Feb 15;8:605393. doi: 10.3389/fmed.2021.605393. eCollection 2021. PMID 33681244

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT03815136/Prot_SAP_001.pdf